CLINICAL TRIAL: NCT06218030
Title: PSIY-744-23: Adjunctive Treatment With L-methylfolate for Treatment-Resistant Generalized Anxiety Disorder: a Pilot Study
Brief Title: Adjunctive Treatment With L-methylfolate for Treatment-Resistant Generalized Anxiety Disorder: a Pilot Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Rafael Freire, Associate Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6038351
Record Dates: First submitted 2023-12-19; First posted 2024-01-23 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder; anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — 5-methyltetrahydrofolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- L-methylfolate arm (Experimental): Oral administration of L-methylfolate 15 mg per day for 8 weeks.
  Interventions: Drug: L-methylfolate

INTERVENTIONS:
Drug: L-methylfolate — Oral administration of L-methylfolate 15 mg per day for 8 weeks. The study drug will be given in addition to the standard of care (SOC) for GAD.

SUMMARY:
The goal of this feasibility study is to determine the tolerability and safety of add on treatment with L-methylfolate in patients with treatment-resistant generalized anxiety disorder (GAD). The primary objective is to monitor for side effects and other risks associated with the treatment. Secondary objectives are to compare the severity of symptoms, serum levels of folate, vitamin B12, C-reactive protein, homocysteine, tumor necrosis factor alpha and interleukin 6 before and after treatment. Participants will continue with their usual treatment for GAD and receive add on treatment with L-methylfolate 15 mg per day for 8 weeks. All participants will receive the same intervention.

DETAILED DESCRIPTION:
Background: Up to 33.7% of the population are affected by an anxiety disorder during their lifetime according to large populationbased surveys. Generalized anxiety disorder (GAD) has a lifetime prevalence of 2.8% to 6.2% in these studies. GAD is associated with functional, occupational, and quality of life impairments. Certain types of medications and psychotherapies are established treatments for GAD, but only 50% of the patients respond to the first treatment trial. Deficiency of folates and neuroinflammation are two hypothesis that could explain why some patients with anxiety disorders do not respond to the usual treatments. Supplementation with folates could correct these deficiencies and reduce inflammation, thus increasing the success rates for treatments. In studies with major depressive disorder, adjunctive folates were associated to higher remission rates. Other studies indicate that folate supplementation lowers homocysteine levels and inflammation. Objectives: Ascertain if adjunctive treatment with Lmethylfolate can produce improvement in treatment-resistant GAD subjects. Methods: This is a proof-of-concept pilot study, an open-label trial of adjunctive treatment with L-methylfolate in patients with treatment-resistant GAD. Ten adult patients with treatment-resistant GAD who have been on a stable dose of an SSRI or SNRI for at least 12 weeks will receive 15 mg doses of L-methylfolate daily for 8 weeks. Patients with moderate to severe major depressive disorder or suicide risk will not be included. Serum levels of folate, vitamin B12, C-reactive protein, homocysteine, tumor necrosis factor alpha and interleukin 6will be measured before and after the trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults.
* Patients on a stable dose of an selective serotonin uptake inhibitors (SSRI) or serotonin and noradrenaline reuptake inhibitors (SNRI) for at least 8 weeks.
* Treatment-resistant GAD, defined by lack of response to at least two drugs, from two different classes of drugs considered first-line or second-line for GAD according to the Canadian Clinical Practice Guidelines for the Management of Anxiety, Posttraumatic Stress and Obsessive-Compulsive Disorders (Katzman et al., 2014). Only trials lasting at least 8 weeks and with at least the minimum effective dose of the given medication will be considered failed trials.

Exclusion Criteria:

* Patients with moderate to severe major depressive disorder based on the Patient Health Questionnaire - Nine Item (PHQ-9) scale (score of 15 or above) at baseline.
* Mini International Neuropsychiatric Interview version (MINI) 7.0 indicates moderate to high current suicidality or "suicide likely in near future" or current suicidal behavior disorder.
* Patients diagnosed with obsessive-compulsive disorder (OCD), bipolar disorder, schizophrenia, schizoaffective disorder, personality disorders, substance use disorders, intellectual disabilities, dementia, epilepsy or other severe neurological diseases.
* Patients with cardiovascular diseases, infections, inflammatory diseases, recent surgeries, recent physical trauma and other medical issues that could produce elevation of c-reactive protein (CRP) or homocysteine.
* Consumption of cannabis, any cannabis by-products, illicit drugs, or alcohol above 3 drinks per week.
* Supplementation of diet with vitamins or consumption of natural health products that may affect anxiety or depression symptoms.
* Reading competence below Grade 5.
* Participants who do not have capacity to conduct consent process.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Throughout the study, 8 weeks
  Monitor participants for treatment-emergent adverse events and serious adverse events.
Incidence of treatment-emergent side effects measured with the ASEC | Baseline visit, 4-week visit and 8-week visit.
  Monitor participants for minor treatment-emergent side effects measured with the Antidepressant Side-Effect Checklist (ASEC).
  ASEC is a list of 21 possible side effects from antidepressants. Each item is rated from 0 (absent) to 3 (severe).
Response to treatment defined by CGI-I score below 3 | 4-week visit and 8-week visit.
  Response to treatment, which will be defined as a score of 1 or 2 on the Clinical Global Impression - Improvement (CGI-I) scale.
  CGI-I is a clinician administered one-item clinical scale rated from 1 (very much improved) to 7 (very much worse). Not assessed would confer score 0.

SECONDARY OUTCOMES:
Remission defined by CGI-S score below 3 | 4-week visit and 8-week visit.
  Remission will be defined as a score of 1 or 2 on the Clinical Global Impression - Severity (CGI-S) scale.
  CGI-S is a clinician administered one-item clinical scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Not assessed would confer score 0.
Change in anxiety severity measured by CGI-S | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for CGI-S by comparing the scores in each visit. CGI-S is a clinician administered one-item clinical scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Not assessed would confer score 0.
Change of anxiety symptoms measured with GAD-7 | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Generalized Anxiety Disorder 7-item scale (GAD-7) by comparing the scores in each visit.
  GAD-7 is a self-rated 7-item scale, each item is rated from 0 (not at all) to 3 (nearly every day).
Change of anxiety symptoms measured with PSWQ | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Penn State Worry Questionnaire (PSWQ) by comparing the scores in each visit.
  PSWQ is a self-rated 16-item scale, each item is rated from 1 (not at all typical of me) to 5 (very typical of me).
Change of anxiety symptoms measured with BAI | Baseline visit, 4-week visit and 8-week visit.
  Changes in scores for Beck Anxiety Inventory (BAI) by comparing the scores in each visit.
  BAI is a self-rated 21-item scale, each item is rated from 0 (not at all) to 3 (severely - it bothered me a lot).
Concentration of CRP in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of C-Reactive Protein (CRP) in serum.
Concentration of homocysteine in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of homocysteine in serum.
Concentration of vitamin B12 in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of vitamin B12 in serum.
Concentration of folate in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of folate in serum.
Concentration of tumor necrosis factor alpha in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of tumor necrosis factor alpha in serum.
Concentration of interleukin 6 in serum | Baseline visit and 8-week visit.
  Collection of blood sample and measurement of the concentration of interleukin 6 in serum.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller AL. The methylation, neurotransmitter, and antioxidant connections between folate and depression. Altern Med Rev. 2008 Sep;13(3):216-26. PMID 18950248
- [Background] Saraswathy KN, Ansari SN, Kaur G, Joshi PC, Chandel S. Association of vitamin B12 mediated hyperhomocysteinemia with depression and anxiety disorder: A cross-sectional study among Bhil indigenous population of India. Clin Nutr ESPEN. 2019 Apr;30:199-203. doi: 10.1016/j.clnesp.2019.01.009. Epub 2019 Feb 12. PMID 30904222
- [Background] Taylor MJ, Carney SM, Goodwin GM, Geddes JR. Folate for depressive disorders: systematic review and meta-analysis of randomized controlled trials. J Psychopharmacol. 2004 Jun;18(2):251-6. doi: 10.1177/0269881104042630. PMID 15260915
- See also: Queen's University Anxiety Research Lab — http://qanxiety.ca